CLINICAL TRIAL: NCT05353179
Title: Phase I, Single-center, Randomized, Double-blind, Single-dose, Parallel Comparison of Pharmacokinetic and Safety Similarities Between Meperizumab Injection and NUCALA® in Healthy Male Volunteers
Brief Title: Study on Pharmacokinetics of Meperizumab Injection and NUCALA® in Healthy Male Volunteers
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TQC3566-I-01
Record Dates: First submitted 2022-04-11; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Granulomatosis With Polyangiitis; Hemophagocytic Syndrome
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Lymphohistiocytosis, Hemophagocytic | interventions — mepolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meperizumab injection (Experimental): Subcutaneous injection of meperizumab once
  Interventions: Drug: Meperizumab injection
- NUCALA® (Active Comparator): Subcutaneous injection of NUCALA® once
  Interventions: Drug: NUCALA®

INTERVENTIONS:
Drug: Meperizumab injection — Meperizumab injection is a humanized monoclonal antibody of IgG1 injection
  Arms: Meperizumab injection
Drug: NUCALA® — NUCALA® is a humanized monoclonal antibody of IgG1 injection
  Arms: NUCALA®

SUMMARY:
The trial was designed as a single-center, randomized, double-blind, single-dose parallel controlled phase I study to evaluate the similarity of pharmacokinetics and safety of Meperizumab injection and NUCALA® in healthy male volunteers.

The plan is to enroll 88 healthy subjects. After signing the written informed consent voluntarily, the subjects will undergo a series of examinations and information collection to determine whether they meet the inclusion criteria. The qualified subjects will be randomized and administered. Biological samples were collected and safety checked before and after administration according to protocol requirements. Adverse events occurred during the trial were collected, and the combination of drug use and non-drug treatment were asked and recorded in detail.

When the 90% confidence interval of geometric mean ratio of the main pharmacokinetic parameters of Meperizumab injection and NUCALA® was within the range of 80.00%-125.00%, it was proved that the pharmacokinetic characteristics of the two were similar.

ELIGIBILITY:
Inclusion Criteria:

* 1 Before the study, the informed consent was signed and the content, process and possible adverse reactions of the test were fully understood;
* 2 Able to complete the research according to the requirements of the test protocol;
* 3 Male subjects aged 18-55 (18 and 55 included);
* 4 Body weight ≥ 50 kg ≤90 kg, body mass index (BMI) ≥ 19 ≤ 26kg/m2;
* 5 Health status: No mental disorders, no history of cardiovascular system, nervous system, respiratory system, digestive system, urinary system, endocrine system and metabolic abnormalities;
* 6 Subjects had no pregnancy plans and voluntarily used effective contraception for at least 6 months from 2 weeks prior to self-medication to their last use of study medication.

Exclusion Criteria:

* 1 Previous neuropsychiatric, respiratory, cardiovascular, digestive, hemolymph, hepatic and renal dysfunction, endocrine, skeletal and musculoskeletal disorders, or other diseases that the investigator judged might affect drug metabolism or safety;
* 2 Known allergy to meperizumab or its excipients;
* 3 Known history of allergic disease or allergy or history of asthma disease;
* 4 Prior treatment with meperizumab or an IL-5 receptor inhibitor, or other antibody or protein drugs that target the IL-5 receptor;
* 5 Who received any live viral vaccines within 2 months prior to infusion of the study drug, or who needed to be vaccinated between the screening period and the end of the study, who used the study drug within 12 months prior to administration of the study drug or planned to receive any monoclonal antibodies or biologic drugs within 12 months after administration of the study drug;
* 6 Patients who have unhealed wounds, ulcers or fractures, or who underwent major surgery within 3 months prior to infusion of the study drug, or who are expected to undergo major surgery within 2 months after study completion;
* 7 Any prescription, over-the-counter, vitamin product or herbal medicine used in the 2 weeks prior to taking the study drug;
* 8 Abnormal and clinically significant examinations during screening period;
* 9 Blood donation or significant blood loss within 3 months prior to taking the study drug (& GT; 450 ml);
* 10 Participated in any drug clinical trials within 3 months prior to taking the study drug;
* 11 Those who smoked more than 5 cigarettes a day 3 months before the experiment;
* 12 History of alcohol abuse (14 units of alcohol per week: 1 unit =360mL beer or 45mL 40% spirits or 150mL wine);
* 13 Those who are screened positive for drugs or have a history of drug abuse in the past five years or have used drugs in the three months prior to the test;
* 14 Screening positive for hepatitis (including hepatitis B and C), acquired immunodeficiency syndrome(AIDS) and syphilis;
* 15 The subject is unable to complete the test due to personal reasons;
* 16 Conditions that other researchers consider inappropriate for inclusion

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Peak concentration(Cmax) | 0 hours before administration (within 60 minutes before administration) to 2016 hours after administration
  Peak maximum plasma drug concentration
Area under drug concentration - time curve(AUC0-t) | 0 hours before administration (within 60 minutes before administration) to 2016 hours after administration
  Area under the curve from zero to the lowest detectable blood drug concentration

SECONDARY OUTCOMES:
The area under the curve extrapolating from zero to infinity(AUC0-∞) | 0 hours before administration (within 60 minutes before administration) to 2016 hours after administration
  Area under the curve from zero to infinity
Peak concentration time(Tmax) | 0 hours before administration (within 60 minutes before administration) to 2016 hours after administration
  Time to reach maximum plasma concentration after dosing
half-life(T1/2) | 0 hours before administration (within 60 minutes before administration) to 2016 hours after administration
  The time it takes for serum drug concentrations to drop by half
Elimination rate constant(λz) | 0 hours before administration (within 60 minutes before administration) to 2016 hours after administration
  The slope of the terminal segment of a semi-logarithmic curve
Residual area percentage(AUC%Extrap) | 0 hours before administration (within 60 minutes before administration) to 2016 hours after administration
  The percentage of the difference between AUC0-∞ and AUC0-t as a percentage of AUC0-t
Apparent clearance(CL/F) | 0 hours before administration (within 60 minutes before administration) to 2016 hours after administration
  Percentage of the body that eliminates organ-scavenging drugs
Apparent volume of distribution(Vd/F) | 0 hours before administration (within 60 minutes before administration) to 2016 hours after administration
  Apparent volume of distribution after non-intravenous administration
Physical examination | 0 hours before administration (within 60 minutes before administration) to 2016 hours after administration
  The doctor will percuss, look, and question the subject, and record any abnormalities in the skin, spine, or limbs
Body temperature | 0 hours before administration (within 60 minutes before administration) to 2016 hours after administration
  Abnormal body temperature
Pulse | 0 hours before administration (within 60 minutes before administration) to 2016 hours after administration
  Abnormal pulse
Blood pressure | 0 hours before administration (within 60 minutes before administration) to 2016 hours after administration
  Abnormal blood pressure
Electrocardiogram(ECG) QT Interval | 0 hours before administration (within 60 minutes before administration) to 2016 hours after administration
  Abnormal ECG QT Interval
Anti-drug antibody(ADA) | 0 hours before administration (within 60 minutes before administration) to 2016 hours after administration
  ADA positive
Neutralizing antibody(NAb) | 0 hours before administration (within 60 minutes before administration) to 2016 hours after administration
  NAb positive

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Changchun University of Traditional Chinese Medicine, Changchun, Jilin, China